CLINICAL TRIAL: NCT02801240
Title: Effect of a Comprehensive Nutrition Support Product on the Nutritional Status of Adults With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Jennifer Ryan, Postdoctoral Fellow, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 031516
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Colitis, Ulcerative; Crohn's Disease
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition Support Product (Experimental): Participants will be asked to take a nutrition support product twice per day for a period of 12 weeks.
  Interventions: Other: Nutrition support product

INTERVENTIONS:
Other: Nutrition support product — Nutrition support product contains macronutrients, micronutrients, phytonutrients, prebiotics, and glutamine. Product is in powder form and is mixed with water or juice before consumption. Taken orally as a nutritional shake twice per day.

SUMMARY:
Individuals with IBD are at risk for nutrient deficiencies. This prospective, non-randomized, open-label study will assess the effect of a nutrition support product on nutritional status in adults with IBD. Up to ten adults with ulcerative colitis or Crohn's disease will be enrolled in the study and asked to take the product for 12 weeks. The primary measures of the study are several blood markers of nutritional status.

DETAILED DESCRIPTION:
It is estimated that 1-1.3 million people in the United States suffer from the Inflammatory Bowel Diseases (IBD) Crohn's disease (CD) and Ulcerative colitis (UC). The pathophysiology of IBD involves malnutrition, malabsorption, altered intestinal permeability, inflammation, and gut flora alterations. Individuals with IBD are at risk for nutrient deficiencies due to decreased intake, decreased absorption and/or increased enteral losses. The most common deficiencies involve many micronutrients including vitamins and minerals; less commonly, adults may also be at risk for macronutrient deficiencies involving protein and total energy intake. The product being studied is a comprehensive nutrition support product that was formulated to meet the nutritional needs of individuals with digestive complaints. This study will assess the effect of the study product on blood markers of nutritional status in adults with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Ulcerative colitis or Crohn's disease (currently active/not considered in remission)
* Willing to have blood drawn twice and willing to fast for 10-12 hours before blood draws
* Able to speak, read and understand English

Exclusion Criteria:

* Currently taking a nutrition support product (macronutrient/micronutrient support product consumed as a reconstituted beverage) or was taken within the last 28 days
* Currently receiving intravenous nutrition support therapy (or within the last 28 days)
* Currently taking curcumin, turmeric, fenugreek, hops, rosemary, ginger or quercetin (or they were taken within the last 14 days)
* Currently taking anti-coagulant or anti-platelet prescription medications (or they were taken within the last 28 days)
* Currently taking antibiotic, antiparasitic, or antifungal medications orally or intravenously (or they were taken within the last 28 days)
* Initiation of or changes to supplements or medications within 28 days prior to screening
* Initiation of or changes to an exercise regimen within 28 days prior to screening
* Initiation of or changes to a food plan within 28 days prior to screening
* Current involvement or within 28 days prior to screening of a significant diet or weight loss program
* Hospitalization (for any reason other than a scheduled medical procedure) within 3 months prior to screening
* Gastrointestinal surgery within 3 months prior to screening
* Currently have a colostomy or ileostomy bag in place
* Malignancy within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
* Women who are lactating, pregnant or planning pregnancy within the next four months
* Difficulty or aversion to taking powdered drink mixes or nutritional shakes
* Currently participating in another interventional research study or participated in another interventional study within the previous 28 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Overall nutritional status | Baseline, 12 weeks
  The effect on overall nutritional status will be determined by aggregating data from multiple measures (albumin, red blood cell count, hemoglobin, hematocrit, vitamin B12, folate, sodium, potassium and calcium) into one reported value. The proportion (percentage) of abnormal values present at baseline will be calculated and compared to the proportion of abnormal values present at the end of the study. Mean change, pre-to-post treatment, will also be assessed for each individual measure.
Albumin, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Red blood cell count | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Hemoglobin | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Hematocrit | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Vitamin B12, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Folate, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Sodium, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Potassium, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.
Calcium, serum | Baseline, 12 weeks
  Mean change, pre-to-post treatment, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Ryan, ND, MS, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No